CLINICAL TRIAL: NCT04330846
Title: Prospective Multicenter Randomized Comparative Study of the Treatment of de Novo Stenosis in Crohn's Disease. Endoscopic Treatment (Self-expanding Metal Prosthesis/Ballon Dilation) vc Surgical Resection (ENDOCIR STUDY)
Brief Title: Prospective Multicenter Randomized Comparative Study of the Treatment of de Novo Stenosis in Chron's Disease.
Acronym: ENDOCIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ENDOCIR
Record Dates: First submitted 2020-03-25; First posted 2020-04-02 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Crohn Disease
Keywords: crohn
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: A prospective multicenter randomized comparative study of the treatment of de novo stenosis due to CD, comparing endoscopic treatment (stent or EBD) vs. surgical resection (SR).
  The type of endoscopic treatment will be initially with EBD and if a failure treatment occurred then a SEMS will be placed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBD group (Experimental): * Post-procedural admission in the Short Stay Unit (SSU).
  * Superficial sedation by endoscopist or anesthesiologist depending on the center.
  * Pneumatic balloon type CRE Boston scientific®; diameter of the balloon at the endoscopist's discretion.
  * A maximum of 2 dilations will be performed with a minimum interval of 15-30 days between each dilation.
  * Dilation failure will be considered if > 2 dilations are required.
  Interventions: Procedure: Surgical resection
- SEMS group (Experimental): * Post-procedural admission in the Short Stay Unit (SSU).
  * Superficial sedation by endoscopist or anesthesiologist depending on the center.
  * Fully coated, self-expanding Tae Woong medical®-type metal prostheses; size of the prostheses at the discretion of the endoscopist
  * Clips can be placed at the distal end of the prosthesis at the endoscopist's discretion.
  * Removal time of the prosthesis 4 weeks.
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Surgical resection — The type of endoscopic treatment will be initially with EBD and if a failure treatment occurred then a SEMS will be placed.

SUMMARY:
Stenosis is one of the most frequent complications in patients with Crohn's disease (CD), causing greater morbidity and increasing the probability of repeated surgery and short bowel syndrome (1-3). Endoscopic balloon dilation (EBD) is clearly the treatment of choice for short stenoses located at the anastomosis of previous surgeries (4-6). However, there is no scientific evidence for determining the most appropriate treatment for de novo stenosis less than 10 cm in length (surgical versus endoscopic treatment), both in terms of efficacy and complications. Neither has it been established which of these two approaches has a greater impact on the quality of life of patients and on costs.

DETAILED DESCRIPTION:
In many cases, a surgical approach allows for the removal of the entire inflamed intestine. However, the percentage of post-surgical recurrence per year after surgery is 80-85% (7), decreasing to 40% in patients who begin preventive immunosuppressive treatment in the immediate post-surgery period (8). This means that more than 40% of patients will require combined immunosuppression to keep CD under control one year after surgery. Endoscopic treatment does not remove the affected intestine. However, it has a long-term therapeutic efficacy of 50-60% with a very low percentage of complications (4-6%).

A large number of studies have shown that patients' quality of life improves when CD is properly controlled, either through medical or surgical treatment (9). However, there are no studies evaluating the quality of life of patients after endoscopic treatment.

Neither are there comparative studies of the costs of the two procedures. However, a recent study comparing the cost of 38 endoscopic procedures with their surgical equivalent suggested that, in most cases, the cost of endoscopic treatment is four times lower (10).

The European Crohn's and Colitis Organization (ECCO) guidelines on the management of de novo stenosis in patients with CD recommend surgery as the first option, based on expert opinion (Level of Evidence 4), although there are no studies comparing the two treatment modalities (11,12).

A Spanish multicenter study coordinated by researchers involved in the present project (Andujar X, et al)(13), which included the largest published series of endoscopic treatment with dilation in patients with CD to date, shows that therapeutic success with EBD in de novo stenoses is achieved in a large percentage of cases, with results similar to those obtained in post-surgical stenoses (73% vs 84%).

In addition, CD stenoses can be treated effectively with self-expanding metal stents (SEMS), and it has been suggested that these may be particularly indicated in patients who are refractory to balloon dilation, including both de novo and anastomotic stenosis patients (14-17). Therefore, in order to compare the efficacy of these two endoscopic treatments, the PROTDILAT study (IP: C Loras. Project FIS nº Pl13/01226 and Clinical Trials. Gov nº NCT02395354) was designed, and is currently in the final manuscript writing phase (100 patients included). The final results (Andújar X, UEGW 2019)(18) confirm that both procedures are effective and safe in the treatment of both post-surgical and de novo stenosis, while showing the therapeutic superiority of EBD over SEMS when the results are evaluated globally (80.5 vs 51.3 %; primary end point). However, this difference is not observed in the subanalysis of patients with stenosis ≥4 cm (LBD: 66.7% vs PMA: 63.6%) but with a significantly lower cost in EDB treatment (EDB 1,212.41 euros vs PMA 3,615.07 euros). Therefore, SEMS may have a role to play in longer stenosis in which EBD has proven to be less efficacious.

This work has been conceived as an exploratory proof of concept study, given that there are currently no studies comparing surgical and endoscopic approaches and it is therefore difficult to calculate the adequate sample size.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age.
* Crohn's disease with predominantly de novo fibrotic stenosis* confirmed by endoscopic and radiological tests, accessible by endoscopy (colonoscopy).
* Patients with known stenosis previously treated with stenting and/or dilation performed over one year before the date of inclusion.
* Symptomatology of intestinal occlusion-subocclusion.
* Refractoriness to conventional medical treatment (non-response to the usual accelerated step-up therapeutic approach).
* Stenosis length < 10 cm.
* Maximum of 2 stenoses.
* Informed consent from patient.

Exclusion Criteria:

* No informed consent from the patient.
* Complicated stenosis with abscess, fistula or significant activity associated with CD not limited to the area of the stenosis.
* Patients with known stenosis previously treated with stenting and/or dilation performed < 1 year before the date of inclusion.
* Pregnancy or lactation.
* Any clinical situation that prevents the performance of endoscopy or surgery.
* Stenosis not accessible by endoscopy.
* Asymptomatic patient.
* Stenosis length ≥ 10 cm.
* Presents with > 2 stenoses.
* Severe coagulation disorders (platelets < 70000; INR > 1.8).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life of patients | One year of follow-up
  Percentage of patients with an increase of more than 30 points in the Inflammatory Bowel Disease Questionnaire (IBDQ-32) quality of life index. The higher the better.

SECONDARY OUTCOMES:
Percentage of patients with clinical recurrence | One year of follow-up
  Percentage of patients with clinical recurrence (scale of obstructive symptoms 0-6) and costs. The lower the better.
Percentage of complications | One year of follow-up
  Percentage of complications and costs.

CONTACTS AND LOCATIONS:
Overall Officials: Carme Loras, Principal Investigator — Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa
Locations (16):
- Spain (16):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Althaia, xarxa assistencial universitaria de Manresa, Manresa, Barcelona
  - Consorci Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Moisès Broggi, Sant Joan Despí, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Cáceres, Cáceres
  - Clínica Girona, Girona
  - Hospital Josep Trueta, Girona
  - Hospital de Inca, Inca
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital de Terrassa, Terrassa
  - Hospital Clínico de Valencia, Valencia
  - Hospital Universitari La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosnes J, Gower-Rousseau C, Seksik P, Cortot A. Epidemiology and natural history of inflammatory bowel diseases. Gastroenterology. 2011 May;140(6):1785-94. doi: 10.1053/j.gastro.2011.01.055. PMID 21530745
- [Background] Solberg IC, Vatn MH, Hoie O, Stray N, Sauar J, Jahnsen J, Moum B, Lygren I; IBSEN Study Group. Clinical course in Crohn's disease: results of a Norwegian population-based ten-year follow-up study. Clin Gastroenterol Hepatol. 2007 Dec;5(12):1430-8. doi: 10.1016/j.cgh.2007.09.002. PMID 18054751
- [Background] Peyrin-Biroulet L, Loftus EV Jr, Colombel JF, Sandborn WJ. The natural history of adult Crohn's disease in population-based cohorts. Am J Gastroenterol. 2010 Feb;105(2):289-97. doi: 10.1038/ajg.2009.579. Epub 2009 Oct 27. PMID 19861953
- [Background] Hassan C, Zullo A, De Francesco V, Ierardi E, Giustini M, Pitidis A, Taggi F, Winn S, Morini S. Systematic review: Endoscopic dilatation in Crohn's disease. Aliment Pharmacol Ther. 2007 Dec;26(11-12):1457-64. doi: 10.1111/j.1365-2036.2007.03532.x. Epub 2007 Sep 28. PMID 17903236
- [Background] Morar PS, Faiz O, Warusavitarne J, Brown S, Cohen R, Hind D, Abercrombie J, Ragunath K, Sanders DS, Arnott I, Wilson G, Bloom S, Arebi N; Crohn's Stricture Study (CroSS) Group. Systematic review with meta-analysis: endoscopic balloon dilatation for Crohn's disease strictures. Aliment Pharmacol Ther. 2015 Nov;42(10):1137-48. doi: 10.1111/apt.13388. Epub 2015 Sep 11. PMID 26358739
- [Background] Navaneethan U, Lourdusamy V, Njei B, Shen B. Endoscopic balloon dilation in the management of strictures in Crohn's disease: a systematic review and meta-analysis of non-randomized trials. Surg Endosc. 2016 Dec;30(12):5434-5443. doi: 10.1007/s00464-016-4902-1. Epub 2016 Apr 28. PMID 27126619
- [Background] Rutgeerts P, Geboes K, Vantrappen G, Beyls J, Kerremans R, Hiele M. Predictability of the postoperative course of Crohn's disease. Gastroenterology. 1990 Oct;99(4):956-63. doi: 10.1016/0016-5085(90)90613-6. PMID 2394349
- [Background] Peyrin-Biroulet L, Deltenre P, Ardizzone S, D'Haens G, Hanauer SB, Herfarth H, Lemann M, Colombel JF. Azathioprine and 6-mercaptopurine for the prevention of postoperative recurrence in Crohn's disease: a meta-analysis. Am J Gastroenterol. 2009 Aug;104(8):2089-96. doi: 10.1038/ajg.2009.301. Epub 2009 Jun 30. PMID 19568226
- [Background] Loras C, Mayor V, Fernandez-Banares F, Esteve M. Study of the standard direct costs of various techniques of advanced endoscopy. Comparison with surgical alternatives. Dig Liver Dis. 2018 Jul;50(7):689-697. doi: 10.1016/j.dld.2018.03.002. Epub 2018 Mar 12. PMID 29610018
- [Background] Wright EK, Kamm MA. Impact of drug therapy and surgery on quality of life in Crohn's disease: a systematic review. Inflamm Bowel Dis. 2015 May;21(5):1187-94. doi: 10.1097/MIB.0000000000000271. PMID 25895008
- [Background] Gionchetti P, Dignass A, Danese S, Magro Dias FJ, Rogler G, Lakatos PL, Adamina M, Ardizzone S, Buskens CJ, Sebastian S, Laureti S, Sampietro GM, Vucelic B, van der Woude CJ, Barreiro-de Acosta M, Maaser C, Portela F, Vavricka SR, Gomollon F; ECCO. 3rd European Evidence-based Consensus on the Diagnosis and Management of Crohn's Disease 2016: Part 2: Surgical Management and Special Situations. J Crohns Colitis. 2017 Feb;11(2):135-149. doi: 10.1093/ecco-jcc/jjw169. Epub 2016 Sep 22. PMID 27660342
- [Background] Bemelman WA, Warusavitarne J, Sampietro GM, Serclova Z, Zmora O, Luglio G, de Buck van Overstraeten A, Burke JP, Buskens CJ, Colombo F, Dias JA, Eliakim R, Elosua T, Gecim IE, Kolacek S, Kierkus J, Kolho KL, Lefevre JH, Millan M, Panis Y, Pinkney T, Russell RK, Shwaartz C, Vaizey C, Yassin N, D'Hoore A. ECCO-ESCP Consensus on Surgery for Crohn's Disease. J Crohns Colitis. 2018 Jan 5;12(1):1-16. doi: 10.1093/ecco-jcc/jjx061. No abstract available. PMID 28498901
- [Background] Andujar X, Loras C, Gonzalez B, Socarras M, Sanchiz V, Bosca M, Domenech E, Calafat M, Rodriguez E, Sicilia B, Calvet X, Barrio J, Guardiola J, Iglesias E, Casanova MJ, Ber Y, Monfort D, Lopez-Sanroman A, Rodriguez-Lago I, Bujanda L, Marquez L, Martin-Arranz MD, Zabana Y, Fernandez-Banares F, Esteve M; ENEIDA registry of GETECCU. Efficacy and safety of endoscopic balloon dilation in inflammatory bowel disease: results of the large multicenter study of the ENEIDA registry. Surg Endosc. 2020 Mar;34(3):1112-1122. doi: 10.1007/s00464-019-06858-z. Epub 2019 May 29. PMID 31144122
- [Background] Attar A, Maunoury V, Vahedi K, Vernier-Massouille G, Vida S, Bulois P, Colombel JF, Bouhnik Y; GETAID. Safety and efficacy of extractible self-expandable metal stents in the treatment of Crohn's disease intestinal strictures: a prospective pilot study. Inflamm Bowel Dis. 2012 Oct;18(10):1849-54. doi: 10.1002/ibd.22844. Epub 2011 Dec 11. PMID 22161935
- [Background] Levine RA, Wasvary H, Kadro O. Endoprosthetic management of refractory ileocolonic anastomotic strictures after resection for Crohn's disease: report of nine-year follow-up and review of the literature. Inflamm Bowel Dis. 2012 Mar;18(3):506-12. doi: 10.1002/ibd.21739. Epub 2011 May 3. PMID 21542067
- [Background] Loras C, Perez-Roldan F, Gornals JB, Barrio J, Igea F, Gonzalez-Huix F, Gonzalez-Carro P, Perez-Miranda M, Espinos JC, Fernandez-Banares F, Esteve M. Endoscopic treatment with self-expanding metal stents for Crohn's disease strictures. Aliment Pharmacol Ther. 2012 Nov;36(9):833-9. doi: 10.1111/apt.12039. PMID 22966851
- [Background] Loras Alastruey C, Andujar Murcia X, Esteve Comas M. The role of stents in the treatment of Crohn's disease strictures. Endosc Int Open. 2016 Mar;4(3):E301-8. doi: 10.1055/s-0042-101786. PMID 27014743
- [Background] Multicenter prospective randomized study to compare endoscopic treatment of strictures in crohn´s disease: self-expanding metal stents vs endoscopic balloon dilation. Protdilat study. Andujar X, Loras Alastruey C, Gornals J.B, Guardiola J., Sanchiz V., Bosca M., Brullet E., Sicília Aladrén B., Naranjo Rodríguez A., Martín-Arranz M.D., Dueñas-Sadornil C., Foruny J.R., Barrio Andrés J., Monfort Miquel D., Busquets Casals D., Pineda J.R., Pérez-Roldán F., Pons Beltrán V., González-Huix Lladó F., Sainz E., Gonzalez B.9,, Reyes Moreno J., Fernández-Bañares F.9,, Esteve M. 27rd United European Gastroenterology Week (UEGW). Barcelona 2019. UNITED EUROPEAN GASTROENTEROLOGY Barcelona 22- 24 October 2019.
- [Derived] Loras C, Ruiz-Ramirez P, Romero J, Andujar X, Bargallo J, Bernardos E, Bosca-Watts MM, Brugiotti C, Brunet E, Busquets D, Cerrillo E, Cortina FJ, Diaz-Milanes JA, Duenas C, Farres R, Golda T, Gonzalez-Huix F, Gornals JB, Guardiola J, Julia D, Lira A, Llao J, Manosa M, Marin I, Millan M, Monfort D, Moro D, Mullerat J, Navarro M, Perez Roldan F, Pijoan E, Pons V, Reyes J, Rufas M, Sainz E, Sanchiz V, Serracant A, Sese E, Soto C, Troya J, Zaragoza N, Tebe C, Paraira M, Sudria-Lopez E, Mayor V, Fernandez-Banares F, Esteve M; Grupo Espanol de Trabajo de la Enfermedad de Crohn y Colitis Ulcerosa GETECCU. Endoscopic treatment (endoscopic balloon dilation/self-expandable metal stent) vs surgical resection for the treatment of de novo stenosis in Crohn's disease (ENDOCIR study): an open-label, multicentre, randomized trial. Trials. 2023 Jun 27;24(1):432. doi: 10.1186/s13063-023-07447-1. PMID 37365665